CLINICAL TRIAL: NCT02682121
Title: Metabolic Alterations in Platelet Study II
Brief Title: Mitochondrial-related Platelet Transcript Expression Levels in Pre-diabetic Subjects Randomized to Metformin or Placebo
Acronym: MAP-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Matthew Rondina, MD, Associate Professor, University of Utah
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1002
Record Dates: First submitted 2015-01-27; First posted 2016-02-15 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Patients on placebo.
  Interventions: Drug: Placebo
- Active drug (Active Comparator): Patients on Metformin, 850mg twice daily for 6mos.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 850 mg twice daily
  Arms: Active drug
Drug: Placebo — Placebo twice daily
  Arms: Placebo

SUMMARY:
Diabetes mellitus (DM) imposes an approximate 2-fold increased risk of atherothrombosis. Patients with type 2 DM have a 2- to 4-fold increase in the risk of coronary artery disease (CAD) and atherothrombotic complications. Current evidence indicates that altered platelet function and "reactivity" are key determinants of arterial and venous thrombosis in metabolic syndromes. In addition, venous thrombosis and pulmonary embolism are associated with increased body mass index, a common feature of type 2 DM and the metabolic syndrome. Altered platelet behavior, function, and phenotype may be critical factors in these thrombotic complications as well. The mechanisms that lead to altered phenotype and function of platelets in DM, and that underlie heightened contributions of platelets to thrombotic complications in type 2 DM, are nevertheless incompletely understood. In this project, the investigators will prospectively determine if clinical intervention with metformin--a commonly-used therapeutic agent that reduces blood glucose, promotes weight loss, and improves lipid profiles--reverses platelet reprogramming and hyperreactivity in obese subjects with impaired fasting glucose and thus, at-risk for type 2 DM.

In addition to metformin, all participants will be given lifestyle modification (LSM) education on diet and physical activity, followed by guidance on how to adhere to the LSM, depending on random assignment to intervention group (education only (n=26) vs. implementation intentions alone (n=27) vs. implementation intentions with partner (n=27)). The LSM coaching for different intervention groups will allow the investigators to test whether there are more effective ways for adherence than others. Participants in these three LSM intervention groups will be further randomized to either Metformin (n=40) or Placebo (n=40), such that participants in the three LSM groups will be randomly and evenly distributed across the two study medication groups.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* BMI>25 kg/m2
* fasting plasma glucose 100-125 mg/dL, AND/OR Hemoglobin-A1C between 5.5 and 6.4%, AND/OR post-load glucose between 140 and 199 mg/dL on a 2-hour Oral Glucose Tolerance Test (OGTT)
* All inclusion criteria will be checked on participants' first in-person visits.

Exclusion Criteria:

* unwilling to accept treatment assignment by randomization
* participation in another clinical research trial
* history of myocardial infarction or stroke
* significant arrhythmia (e.g. atrial fibrillation)
* active thromboembolic disease
* inflammatory bowel disease
* serum creatinine levels greater than or equal to 1.5 mg/dL in males or greater than or equal to 1.4 mg/dL in females
* known hypersensitivity to metformin hydrochloride or any of its components
* acute or chronic metabolic acidosis
* inability to participate in lifestyle modifications
* pregnancy; other glucose-lowering or diabetic therapy
* systemic glucocorticoids
* prescription weight loss medications
* or otherwise deemed unsuitable by study investigators (e.g. unable to complete follow-up visits, alcohol abuse, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be gene expression levels of mitofusin 2 and uncoupling protein 2 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Weyrich, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States